CLINICAL TRIAL: NCT06354426
Title: Short-term Mortality and Readmission Rate Prediction by the Sequential Organ Failure Assessment Score in Acute Decompensated Heart Failure
Brief Title: Short-term Mortality Prediction by the SOFA Score in Acute Decompensated Heart Failure
Status: Completed | Type: Observational
Sponsor: Hanoi Heart Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: BVT2022/01
Record Dates: First submitted 2024-03-30; First posted 2024-04-09 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Acute Decompensated Heart Failure
Keywords: SOFA score; Acute decompensated heart failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data on the use of sequential organ failure assessment (SOFA) in patients with cardiovascular disease are increasing. Several studies demonstrated that the SOFA score can identify short-term mortality in patients with acute decompensated heart failure (ADHF). This study was conducted to determine the prognostic value of the admission SOFA score in patients hospitalised for ADHF and to assess its ability in predicting the 30-day readmission rate.

ELIGIBILITY:
Inclusion Criteria:

* All patients over 18 years old who were hospitalised for acute heart failure were included (either new-onset acute heart failure or ADHF).

Exclusion Criteria:

* Patients with septic shock or pulmonary infarction were excluded.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: This was a single-centre, prospective study conducted from July 2022 to August 2023 at Hanoi Heart Hospital (Hanoi, Vietnam).
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Mortality | Within 30 days from the day of hospitalization
  The sequential organ failure assessment (SOFA) score was used to assess the relation to the all cause mortality of the patient with acute decompensated heart failure. Higher SOFA score is correlated with higher in-hospital mortality rate and 30-day mortality regardless of age, gender, or other comorbidities.

SECONDARY OUTCOMES:
Re-admission rate | Within 30 days
  To assess the prediction ability of the sequential organ failure assessment (SOFA) score in regard of re-admission rate.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Heart Hospital, Hanoi, Hoan Kiem, Vietnam